CLINICAL TRIAL: NCT05371626
Title: Suture-less Procedure for Management of Cicatricial Upper Eyelid Entropion
Brief Title: Cicatricial Upper Eyelid Entropion Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farag Khalil Ibrahiem, Assistant Professor, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oculoplastic clinic
Record Dates: First submitted 2022-05-05; First posted 2022-05-12 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Entropion
MeSH Terms: conditions — Entropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suture-less entropion technique (Other): suture-less technique for cicatricial entropion
  Interventions: Procedure: Suture-less surgical procedure

INTERVENTIONS:
Procedure: Suture-less surgical procedure — Suture-less technique will be used in treatment for cicatricial upper eyelid entropion

SUMMARY:
Suture-less technique will be used in treatment for cicatricial upper eyelid entropion to detect its long-term efficacy

ELIGIBILITY:
Inclusion Criteria:

* Upper eyelid cicatricial entropion with no history of previous surgery.
* Cooperative patients older then 16 years old.

Exclusion Criteria:

* Previous lid surgery.
* Senile and mechanical entropion.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Eyelid margin reposition to the normal position | 1 month
  posterior edge of eyelid opposed to eye globe using slit lamp examination of the inner margin of the upper lid

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided